CLINICAL TRIAL: NCT00133523
Title: Comparative Study of Influenza Vaccines in Adults - FLU-VACS
Brief Title: FLU-VACS Comparative Study in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-060; IRBMed# 2004-0334
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2009-10

CONDITIONS: Influenza
Keywords: FLU-VACS, influenza, vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group 4: Placebo: Intramuscular (Placebo Comparator): N=165 subjects administered placebo intramuscularly.
  Interventions: Other: Placebo
- Group 3: Placebo: Nasal (Placebo Comparator): N=165 subjects administered placebo intranasally.
  Interventions: Other: Placebo
- Group 1: FluMist™ (Experimental): N=825 subjects administered live attenuated vaccine intranasally.
  Interventions: Biological: Cold-adapted live attenuated influenza virus vaccine, trivalent
- Group 2: Fluzone®/Fluvirin (Experimental): N=825 subjects administered inactivated vaccine intramuscularly.
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Cold-adapted live attenuated influenza virus vaccine, trivalent — Live-attenuated influenza vaccine; single annual dose administered as an intranasal spray.
  Arms: Group 1: FluMist™
Other: Placebo — Physiological saline administered as an intramuscular injection.
  Arms: Group 4: Placebo: Intramuscular
Biological: Trivalent inactivated influenza vaccine — Inactivated influenza vaccine; single annual dose administered as an intramuscular injection..
  Arms: Group 2: Fluzone®/Fluvirin
Biological: Trivalent inactivated influenza vaccine — Inactivated influenza vaccine; single annual dose administered as an intramuscular injection.
  Arms: Group 2: Fluzone®/Fluvirin
Other: Placebo — Normal allantoic fluid administered annually as an internasal spray.
  Arms: Group 3: Placebo: Nasal

SUMMARY:
The purpose of this study is to compare 2 licensed flu vaccines to each other and to placebo (inactive substance). The study will be conducted among healthy adult participants aged 18-49 years and is expected to last 3 years. During year 1, participants will be assigned to receive 1 of the 2 licensed flu vaccines or placebo, given as either nasal spray (live-attenuated vaccine or placebo) or injection (inactivated vaccine or placebo). Participants will receive the same assigned vaccine or placebo during year 2. During year 3, participants will be followed, but will not receive flu vaccine. Each year blood samples will be collected before and 1 month after each vaccination and at the end of each flu season in order to measure how the body responds to the vaccine and how well participants were protected from the flu. During the flu season, participants with flu-like illness will provide information on symptoms and provide a throat swab to test for virus identification.

DETAILED DESCRIPTION:
Influenza occurs on an annual basis, producing significant mortality in most years, mainly in those with underlying conditions and those at extremes of age. This study is a placebo-controlled trial to examine efficacies of the live attenuated and inactivated influenza vaccines, and immune correlates of protection; the study will take place in Michigan over a three year period, and will target adults aged 18-49 years. Both vaccine preparations are licensed for this age group. In the first year, participants will be randomly assigned to receive one of the two licensed vaccines or placebo. In the second year, participant receipt of vaccine (updated according to national recommendations) or placebo will continue as assigned in the first year for returning participants, and new enrollees will be randomly assigned to intervention. In the third year, when duration of immunity will be evaluated, no interventions will be given. In all study years, blood specimens for serologic studies and specimens for virus identification will be collected and a number of laboratory studies will be performed so that it will be possible to achieve the study's objectives. The primary annual study outcome for efficacy is the proportion of subjects with laboratory-confirmed symptomatic influenza A or B illness, defined as influenza virus isolated in tissue culture from a throat swab obtained from a participant during an episode of illness meeting the influenza case definition that is confirmed as influenza by fluorescent antibody or polymerase chain reaction (PCR) techniques; or serologic confirmation of influenza infection in a participant with an episode of illness meeting the influenza case definition, specifically a 4-fold rise in hemagglutinin inhibition assay (HAI) antibody titer to a circulating influenza strain between post-vaccination (pre-season) and post-season paired sera. The influenza case definition is illness with at least one respiratory symptom (cough or nasal congestion) and at least one constitutional symptom (fever or feverishness, chills or body aches). Subjects will be evaluated for serious adverse events throughout each annual study period. Annually, the proportion of participants with local reactions during the first seven days or any adverse reactions during the first thirty days after vaccine receipt will be compared with recipients of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Persons must be adult men and women aged 18-49 years.
* Persons must be able and willing to provide informed consent.
* Persons must expect to reside in the study area during the entire study period and be interested in participating each year.
* Persons must be willing to receive the licensed live-attenuated vaccine (FluMist) or placebo given as a nasal spray, or the licensed inactivated influenza vaccine (Fluzone or Fluvirin) or placebo given as an intramuscular injection.
* Persons must be willing to provide multiple blood specimens collected by venipuncture each year they are in the study. During each of the first two years of study, blood specimens will be collected three times - at the enrollment visit (immediately prior to administration of vaccine or placebo), at the first follow-up visit 3-5 weeks later, and at the end of the influenza season visit (approximately 4-6 months later); during the third year of the study, blood specimens will be collected twice only, at visits before and after the influenza season.
* Persons must be willing to notify study personnel in the event of influenza-like illness, to provide information on illness symptoms, and to permit collection of a throat culture (swab) specimen for laboratory studies.
* Persons must be willing to not receive an influenza vaccine while participating - other than that (influenza vaccine or placebo) received as study medication.

Exclusion Criteria:

* Persons with any health condition for which the inactivated vaccine is recommended (Advisory Committee on Immunization Practices - ACIP) including: chronic diseases of the pulmonary or cardiovascular systems (including asthma); chronic metabolic diseases (including diabetes); renal dysfunction; hemoglobinopathies; immune deficiency disease (including HIV infection) or on-going immunosuppressive therapy.
* Persons who are currently pregnant, nursing mothers or planning a pregnancy within one month of vaccination.
* Persons with hypersensitivity to egg, egg protein, thimerosal (a preservative) or the antibiotic Gentamicin (also know as Garamycin).
* Persons who have had a prior serious reaction to influenza vaccine, or ever had Guillain-Barre syndrome.
* Persons who are living in a household with or have direction occupational contact with immunosuppressed individuals (including health care workers with direct patient contact).
* Persons who have received an influenza vaccine for the influenza season in which they are to be first enrolled or those who plan to receive an influenza vaccine during their participation in the study - other than that (influenza vaccine or placebo) received as study medication.
* Persons who have received any other vaccine within one week prior to enrollment (may delay enrollment).
* Persons who have had a respiratory illness or illness with fever within 3 days of study enrollment (may delay enrollment).
* Persons who are participating in another research study involving any study medications (medicines or vaccines).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2349 (Actual)
Dates: Start 2004-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The appearance among patients of symptomatic laboratory-confirmed influenza. | Influenza season Nov-Apr. Within 72 hours of illness onset throat swab specimens will be obtained from participants with influenza like illness (ILI).

SECONDARY OUTCOMES:
Any measurable increase in antibody titers, and the proportion with antibody levels considered protective. | Annual enrollment, post vaccination Oct-Jan, and post season Apr-May.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ann Arbor West, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Western Michigan University Health Services, Kalamazoo, Michigan
  - Livonia East, Livonia, Michigan
  - Central Michigan University Health Services, Mount Pleasant, Michigan
  - Eastern Michigan University Health Services, Ypsilanti, Michigan

REFERENCES:
- [Result] Ohmit SE, Victor JC, Rotthoff JR, Teich ER, Truscon RK, Baum LL, Rangarajan B, Newton DW, Boulton ML, Monto AS. Prevention of antigenically drifted influenza by inactivated and live attenuated vaccines. N Engl J Med. 2006 Dec 14;355(24):2513-22. doi: 10.1056/NEJMoa061850. PMID 17167134
- [Result] Ohmit SE, Victor JC, Teich ER, Truscon RK, Rotthoff JR, Newton DW, Campbell SA, Boulton ML, Monto AS. Prevention of symptomatic seasonal influenza in 2005-2006 by inactivated and live attenuated vaccines. J Infect Dis. 2008 Aug 1;198(3):312-7. doi: 10.1086/589885. PMID 18522501
- [Derived] Petrie JG, Ohmit SE, Johnson E, Cross RT, Monto AS. Efficacy studies of influenza vaccines: effect of end points used and characteristics of vaccine failures. J Infect Dis. 2011 May 1;203(9):1309-15. doi: 10.1093/infdis/jir015. Epub 2011 Mar 4. PMID 21378375